CLINICAL TRIAL: NCT04387487
Title: Effect of Multimedia Video Information in Relieving Anxiety Related to Spinalanesthesia. A Randomized Control Trial
Brief Title: Does Showing Video Information About Spinal Anesthesia Relieves Patient Anxiety?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chitwan Medical College (Other)
Responsible Party: Principal Investigator, Dr Deepak Bhandari, Consultant Anesthesiologist, Chitwan Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMC001
Record Dates: First submitted 2020-04-30; First posted 2020-05-13 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Anxiety; Surgery; Spinal Anesthesia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Intervention name- multimedia video information Intervention details- multimedia video information of 4.5 mins regarding procedure, indication and complications related to spinal anesthesia will be shown to patients in intervention group , patient will be allowed to ask questions.
Who Masked: Participant, Investigator
Masking Description: participant and investigators will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Group (Experimental): Video Group
  multimedia video information of 4.5 mins regarding procedure, indication and complications related to spinal anesthesia will be shown to patients in intervention group , patient will be allowed to ask questions.
  Interventions: Behavioral: Multimedia video information
- non video group (No Intervention): patients in control group will be given verbal information regarding procedure, indication and complication, patient will be allowed to ask questions.

INTERVENTIONS:
Behavioral: Multimedia video information — During pre anesthesia visit after regular pre anesthesia check up patient will be asked to fill the Hamilton scoring questionnaire about anxiety.
  After this a multimedia video information about spinal anesthesia of around 6 minutes will be shown to the intervention group during pre anesthesia visit. This video will contain explanation about how spinal anesthesia procedure is conducted. Patient will be allowed to ask questions.
  On the day of surgery in the pre surgical area again Hamilton scoring questionnaire will be asked with the patients to check the level of anxiety.
  Arms: Video Group

SUMMARY:
Our primary aim is to compare the effect of pre-operative multimedia video information on perioperative anxiety and hemodynamic parameters.

DETAILED DESCRIPTION:
Anxiety is common in perioperative patients with incidence of 60-89 %. Lack of knowledge about surgery and anesthesia, anesthesia procedures and unfamiliar surroundings are the common causes of anxiety . Anxiety related to anesthesia can be due to lack of knowledge about its process, procedures and risk associated with it or misconceptions about it. Long NPO status and unexpected delay before and during anesthesia procedure and surgery further increases the anxiety in perioperative patients. Anxiety increases the activity of sympathetic nervous system and cause preoperative and intraoperative tachycardia, hypertension, arrhythmias, increased pain perception and increase requirement of anaesthetic drugs. This may lead to harmful effect on patient health and decrease overall patient satisfaction and even traumatic experience for rest of life. This may affect process of giving informed consent for the planned surgery. Many measures are taken to allay anxiety in perioperative patients. Anxiolytic medications are given preoperative period to allay anxiety but they may have detrimental effect on patient health, requires administration under supervision of health professional and may not be effective unless the cause of anxiety is taken care. Counselling regarding the procedure of anesthesia during pre-anesthetic check up is other way to allay anxiety but transfer of knowledge is usually limited and may not be entirely retained. Other method in the form of written pamphlets, booklet or questionnaires have been tried but most of the patients in Nepal are not literate enough to read and understand it. Multimedia information to allay patient's anxiety has been successfully tried. Previous study shows a significant reduction in anxiety level due to preoperative multimedia information among the patients undergoing surgery. Investigators have developed a short visual clip of 4.5 minutes duration depicting the procedure of spinal anaesthesia .Investigators will be using Hamilton Anxiety Score in patients undergoing surgical procedures under spinal anesthesia .

ELIGIBILITY:
Inclusion Criteria:

- All patients between 18 and 65 years of age of either sex undergoing elective surgery under SAB were included.Only patients in ASA category 1 and 2 will be included.

Exclusion Criteria:

* Patients refusing to give consent for the study,

  * Patients Having significant cardiovascular or neurological disease,
  * Patients On medications such as beta blockers, antidepressants, cardiac or psychiatric drugs,
  * Pregnant patients and
  * Patients those who had undergone procedures under SAB in the past
  * Patients facing any major complications after the surgery such as massive blood loss, having to convert to general anesthesia due to lengthy surgical procedure, patients requiring critical care administration after the surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-05 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety | 1) During pre anesthesia check up before providing verbal or multimedia information. 2) one hour before the surgery 3) 8 hours after the surgery
  1. During pre anesthesia visit before conduction pre anesthesia checkup a base line level anxiety will be measured among both the group of patients.
     After this pre anesthesia examination will be conducted. The intervention group will be then asked to watch multimedia video information where as other group will be provided with verbal information only.
  2. Change in anxiety level will be measured at one hour before the surgery and eight hours after the surgery among the both the group using same scoring system.
  Change in anxiety level will be assessed using the Hamilton anxiety rating scale which ranges from minimum 0 and maximum 56 (higher score means poor outcome high level of anxiety)

IPD SHARING:
Plan to Share IPD: Yes
patients Hamilton scores and data regarding the study will be provided.
Supporting Information: Study Protocol, ICF
Time Frame: data will be available after the study is completed to only people who request to view the data
Access Criteria: data will be shared only for academic purpose

REFERENCES:
- [Background] Hashimoto Y, Baba S, Koh H, Takagi H, Ishihara H, Matsuki A. [Anxiolytic effect of preoperative showing of "anesthesia video" for surgical patients]. Masui. 1993 Apr;42(4):611-6. Japanese. PMID 8315804